CLINICAL TRIAL: NCT03250780
Title: Chromoendoscopy With 0.03% Indigo-carmine Delivered Via a Foot Pump Compared With 0.2% Indigo-carmine Delivered Via Spray Catheter for Detecting Dysplasia in Patients Undergoing Surveillance in Inflammatory Bowel Disease. A Randomized Control Trial.
Brief Title: Chromoendoscopy in Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GA16/89362
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Indigo Carmine

ARMS (1):
- Patients with extensive colitis (Experimental): Patients with extensive colitis, for at least 8-10 years, already on the surveillance programme or newly referred whilst attending their outpatients IBD clinic at Leeds Teaching Hospitals NHS Trust will be screened by one of the research doctors who will be performing the surveillance colonoscopy.
  Interventions: Procedure: indigo-carmine 0.2% using a spray catheter; Procedure: 0.03% using a foot pump

INTERVENTIONS:
Procedure: indigo-carmine 0.2% using a spray catheter
Procedure: 0.03% using a foot pump

SUMMARY:
Patients with longstanding ulcerative colitis (inflammatory bowel disease, IBD) have increased risk of developing colorectal cancer (CRC) when compared with that of the general population. Therefore patients with longstanding colitis undergo regular screening colonoscopy at varied time intervals depending on their individual risk. This is thought to detect early mucosal (interior bowel lining) abnormalities, known as dysplasia, which can progress to CRC. Until recently, IBD surveillance has relied upon colonoscopy with multiple (at least 33) random biopsies of the bowel lining to detect dysplasia, but now international guidelines recommended a technique called chromoendoscopy.

Chromoendoscopy involves applying a dye, called indigo-carmine, to the bowel lining whilst performing colonoscopy which highlights more subtle abnormalities, therefore increasing dysplasia detection rate.

There is no standard international concentration of the dye spray used during chromoendoscopy. Studies have used different concentrations of indigo-carmine dye ranging from 0.1 to 0.4%. We have recently shown that 0.2% dye improves detection rates compared to high definition white light. The recent international SCENIC guidelines suggest using 0.03% indigo-carmine via a foot pump. However there are no trials comparing the two methods and no previous trials have used the 0.03%. We therefore aim to perform a randomised control trial, comparing 0.03% indigo-carmine dye versus 0.2% in detecting dysplasia in patients undergoing surveillance colonoscopy in IBD. Any lesions seen will assessed using standard endoscopic appearance but also using optical biopsy forceps to further characterise the lesion, then manage the lesion as standard guidelines. We will also take two additional rectal biopsies, which will be snap frozen in liquid nitrogen and then studied using Raman Spectroscopy, Infra Red spectroscopy and electrochemical impedance to develop optical markers to identify patients at higher risk of dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with longstanding (more than 8 years of disease), extensive (extending proximal to splenic flexure) colitis attending for surveillance colonoscopy. 2) Patients aged over 18 years of age 3) Patients with Primary Sclerosing Cholangitis and Inflammatory Bowel Disease colitis.

Exclusion Criteria:

* 1) Pregnant 2) Unwilling or unable to give informed consent 3) Severe active colitis 4) Poor bowel preparation 5) Unable to reach the caecum

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least low grade dysplasia detected by targeted biopsy using 0.2% indigo-carmine compared with 0.03% indigo-carmine. | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom